CLINICAL TRIAL: NCT06904937
Title: Renal Manifestations During Idiopathic Inflammatory Myopathies: Real-life Study of an Alsatian Cohort (France)
Brief Title: Renal Manifestations During Idiopathic Inflammatory Myopathies
Acronym: IIM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9136
Record Dates: First submitted 2024-07-05; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Myopathy
Keywords: Inflammatory Myopathy; Idiopathic Inflammatory Myopathy; Renal biopsy,; Guided kidney aspiration biopsy
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are currently no recommendations regarding treatments for Idiopathic Inflammatory Myopathies (IIM) due to the difficulty in conducting high-powered randomized controlled trials.

Generally speaking, corticosteroids constitute one of the cornerstones of treatment and are, with some exceptions, always used at least in the initial phase of the disease. In general, this involves oral corticosteroid therapy initiated between 0.5 and 1.5 mg/kg/day followed by a gradual decrease after 4 to 6 weeks of treatment. It is generally necessary to introduce immunosuppressive treatment early with the aim of avoiding corticosteroids. The most commonly used as first-line treatment and having shown effectiveness in observational studies are methotrexate, azathioprine, mycophenolate mofetil and calcineurin inhibitors. In general, rituximab is reserved for severe forms refractory to several first-line immunosuppressants, and has shown some effectiveness during a randomized study. Likewise, cyclophosphamide is only considered in the most severe forms, generally rapidly progressive interstitial lung damage. More recently, Janus kinase inhibitors have been evaluated in several open-label and small-number studies, showing interesting effectiveness, particularly for refractory forms, as shown in this recent review of the literature. Immunoglobulins are the only treatment that has shown superiority compared to placebo in good quality randomized controlled studies. However, due to their cost and difficulty of access, they should be reserved for the severe form, particularly in cases of dysphagia, or refractory form.

Apart from these medicinal treatments, it is necessary to add all the non-drug measures which are an integral part of the management of IIM. Performing regular physical activity helps prevent muscle loss and also has a beneficial effect on other comorbidities often present in patients and aggravated by corticosteroid therapy, such as cardiovascular risk factors, osteoporosis and resistance to 'insulin.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 18 years old)
* Inflammatory myopathy defined by the ACR/EULAR 2017 criteria
* Kidney biopsy performed
* Supported at the Strasbourg University Hospital during the period from January 1, 1990 to May 1, 2023.
* Subject who has not expressed opposition to the reuse of their data for scientific research purposes.

It is the responsibility of the investigator to verify the absence of opposition in the patient's medical file.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Known etiology of renal damage excluding inflammatory myopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) having inflammatory myopathy and hospitalized at the Strasbourg University Hospital during the period from January 1, 1990 to May 1, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Describe the characteristics of patients with inflammatory myopathies | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie - CHU de Strasbourg - France, Strasbourg, France